CLINICAL TRIAL: NCT00644618
Title: Randomized Controlled Trial of Gemcitabine Combined With 125I Brachytherapy Versus Gemcitabine Alone in Patients With Locally Advanced Pancreatic Cancer
Brief Title: Randomized Controlled Trial of Gemcitabine Combined With 125I Brachytherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: President Hu Yu, Union hospital, Huazhong University of Science and Technology
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Union Hospital
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Locally Advanced Pancreatic Cancer
Keywords: pancreatic cancer; locally advanced
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: gemcitabine
- B (Experimental)
  Interventions: Other: 125I brachytherapy PLUS gemcitabine

INTERVENTIONS:
Drug: gemcitabine — a 30-minute intravenous infusions of gemcitabine 1,000 mg/m2 weekly×7, followed by a 1-week pause, and then weekly×3
  Arms: A
Other: 125I brachytherapy PLUS gemcitabine — 125I brachytherapy PLUS a 30-minute intravenous infusions of gemcitabine 1,000 mg/m2 weekly×7, followed by a 1-week pause, and then weekly×3
  Arms: B

SUMMARY:
For patients with unresectable locally advanced pancreatic cancer, the combined use of external-beam radiation therapy (EBRT) and systemic chemotherapy of 5-FU has been widely recognized as the most effective chemoradiotherapy approach.But most patients succumb to local recurrence and metastasis after treatment, and the prognosis remains poor On the basis of the development and superiority of the interstitial brachytherapy and the radiosensitizing effect of gemcitabine, we performed a clinical study to explore the interaction of improved I-125 brachytherapy and gemcitabine and compare the regimen to the standard gemcitabine treatment specifically in patients with non-metastatic, unresectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven
* locally advanced pancreatic adenocarcinoma stage
* No systemic metastases
* Age between 18-75
* Karnofsky-Performance Status equal to, or greater than 70 %
* At least a 2-dimensionally measurable tumor lesion
* Adequate renal and liver function
* Written consent statement
* Patients' compliance and geographical proximity
* Life expectancy equal to or greater than 3 months

Exclusion Criteria:

* Serious psychological disease
* Pregnancy and inadequate or not secure contraception or breastfeeding women
* Other previous malignant disease in the past two years
* Serious systemic concomitant diseases, excluding participation in a trial
* Other experimental treatment during or within 6 weeks prior to this trial (including chemotherapeutic medicine or immune-therapies)
* Every other condition or therapy assessed by the physician as an eventual risk for the patient or restricting the aims of the trial
* Distant metastasis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2003-01; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Survival | 2 years after the inclusion of the last patient

SECONDARY OUTCOMES:
response rate, clinical benefit response, and safety | 2 month after the treatment finished